CLINICAL TRIAL: NCT00043641
Title: HIV Expression in Patients With Viral Loads Suppressed on HAART
Brief Title: HIV Expression in Patients With Low Viral Load on Highly Active Antiretroviral Therapy (HAART)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020232; 02-I-0232
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2013-02-07

CONDITIONS: HIV Infections
Keywords: RT PCR; Antiretrovial Therapy; Drug Intensification; Ultra-low; Sequence; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

SUMMARY:
This study will investigate low-level viral loads in HIV-infected patients taking highly active antiretroviral therapy (HAART). Although HAART reduces viral levels and restores immune function to some degree, it does not cure HIV infection. The virus persists even at levels below that which it can be detected. This study will examine where this residual virus comes from in order to better understand the infection and the effectiveness of therapies. In addition, the study will 1) evaluate the ability of a new test to detect the virus at low levels; and 2) determine whether adding the protease inhibitor Kaletra to the HAART treatment regimen for patients with a low viral load will further decrease their viral load.

HIV-infected patients 18 years of age and older may be eligible for this study. Patients involved in the viral load test will be recruited from an NIAID HIV study in which they are already participating. Three groups of patients will be enrolled: those with a viral load of less than 50 copies/ml plasma, those with 51-500 copies/ml, and those with 501-5000 copies/ml. Patients involved in the Kaletra trial must have been taking HAART for 6 months or more and have less than 50 viral copies/ml plasma. They will be screened for this study with a history, physical examination, and routine laboratory tests.

Participants in the viral load test evaluation will donate 70 ml of blood up to four times. No more than one sample will be collected per day.

Participants in the Kaletra trial will have blood samples drawn on two successive days and will then be randomly assigned to one of two treatment groups. One group will begin Kaletra therapy (four capsules two times a day) immediately; the other will undergo observation for 4 weeks before starting Kaletra. Depending on what group they are in, patients will provide blood samples for viral load measurements and clinical samples according to the following schedule:

Immediate Kaletra

One sample each during weeks 1, 2, and 3, of therapy and two samples during week 4.

Delayed Kaletra

One sample each during weeks 1, 2, and 3 of observation and two samples during week 4. After starting therapy, one sample will be collected each week during weeks 1, 2, and 3 of therapy and two samples during week 4.

In both groups, after the last dose of medicine on day 28, Kaletra therapy will be complete. At the end of therapy, additional blood will be collected for viral sampling as follows: one sample each during weeks 1, 2, and 3, and two samples during week 4 after Kaletra therapy.

DETAILED DESCRIPTION:
This protocol is an exploratory study of HIV expression in patients who are receiving highly active antiviral therapy and who have low viral loads below or near the current limit of detection (50 copies/ml plasma). Recent studies have suggested that patients with suppressed viral loads in this low range have continued HIV expression, but the amount and the origin of this virus remains unknown. The amount of virus expression in plasma is uncertain because the current viral load assays are imprecise in the cutoff range of 50-75 copies/ml plasma. The origin of the HIV found at low viral loads detected is unknown as well; two possible sources of virus include expression from long-lived reservoirs of infected cells, and low level spreading infection to uninfected cells. Determining the origin of HIV expression has clinical importance; currently available HIV drug therapy will have little effect on HIV expression from established reservoirs, but more potent HIV therapy could potentially inhibit a spreading HIV infection.

In this study we plan two principal objectives. First, we will investigate the level of HIV expression in plasma samples at low viral loads using a new HIV load assay with enhanced sensitivity and precision in the viral load range of 1-100 copies. If data from the survey confirms acceptable performance characteristics for this assay we will proceed with stage II of the protocol. In stage II we plan to determine, in several short-term intensification approaches to investigate whether the incorporation of an additional antiretroviral to suppressive HAART regimens ("intensification HAART") will further suppress plasma virus. In a small pilot study, we will plan to intensify regimens for 30 days in a nonrandomized fashion. Secondly, we plan to study patients who are switching medications for preference or mild toxicity. In these patients we will intensify their regimens for 30 days in an overlap fashion, adding the new drug instead of switching medications. After 30 days of drug overlap, we will continue the new drug and discontinue the identified antiretroviral. These initial studies will assist in obtaining initial data and confirming the estimated sample size of a larger, randomized study to rigorously investigate the virologic effects of drug intensification. If these initial proof-of-concept experiments suggest that HIV may be suppressed by intensification HAART, then we plan to expand the study in a larger controlled trial to determine the degree of suppression possible with intensification therapy.

As a secondary objective we will investigate whether it is feasible to study HIV genetic variation in samples from patients with suppressed viral loads using molecular techniques developed to study HIV variation in patients with viral loads greater than 1000 copies/ml plasma (protocol 00-I-0110).

We plan to enroll up to 70 patients in a viral load survey cohort of HIV viral loads, and analyze a series of samples from completed trials of antiretroviral therapy.

ELIGIBILITY:
* INCLUSION CRITERIA: VIRAL SURVEY COHORT
* HIV-1 infection documented by HIV ELISA and WB
* Age greater than or equal to 18 years old
* Hemoglobin greater than or equal to 12 mg/dl within the last six weeks
* On HAART according to current DHHS guidelines.
* Most recent viral load (within the last 12 weeks):

  * less than 50 by bDNA or RT-PCR (65 patients)
  * 50-500 by bDNA or RT-PCR (3 patients)
  * 501 - 10,000 by bDNA or RT-PCR (2 patients)

EXCLUSION CRITERIA:

-Any febrile illness (T greater than 38.0 degrees C) in the 3 weeks prior to blood draw.

VIRAL SURVEY COHORT- M98-863, M97-720, AACTG 5201 SAMPLES (no inclusion/exclusion):

-Samples from patients enrolled in the completed M98-863, M97-720 or AACTG 5201 study.

INCLUSION CRITERIA: PILOT INTENSIFICATION COHORT:

* HIV-1 infection documented by HIV ELISA and WB
* Age greater than or equal to 18 years old
* Hgb greater than or equal to 12 mg/dl
* CD4 greater than 200 cells/ micro liter and CD4% greater than 14% and not requiring prophylaxis for opportunistic infections
* Therapy with accept HAART regimen for greater than or equal to 6 months
* Viral load less than 50 copies RNA/ml plasma by RT-PCR for at least four months
* Viral load greater than 0.38 copies RNA/ml plasma by SCA assay or positive in the adapted Amplicor assay
* Current HAART with DHHS-approved regimen NRTI+PI, NRTI alone, NRTI+NNRTI.
* Willingness to take an additional antiretroviral to current regimen for 30 days.
* For patients to start lopinavir/ritonavir, willingness to reduce the dose of sildenafil and other co-administered medicines that may be affected by the addition of lopinavir/ritonavir during the course of therapy with lopinavir/ritonavir
* For patients to start efavirenz arm, willingness to take efavirenz and adjust other medications or supplements as necessary, and to be aware that efavirenz is contraindicated in pregnancy and that may result in false positive urine tests for THC
* For patients starting raltegravir, no prior history of rhabdomyolysis and no co-administration of agents which, in the opinion of the investigators, would cause rhabodomyolysis or myopathy.
* Patient must have primary care outside this protocol.
* Patients must practice accepted barrier methods to prevent pregnancy.
* For patients enrolled in piolt study of suppression after development of resistance, patient must have documented evidence of prior drug resistance either: Prior resisteance testing with the presence of resisnce mutations or documents evidence of viral RNA levels greater than 100 copies/ml plasma for greater than 6 months despite antiretroviral thereapy. Patients with prior therapy on monotherapy or suboptimal combination therapy ARE eligible for this study.

INCLUSION CRITERIA: RANDOMIZED INTENSIFICATION COHORT (NIH, University of Pittsburgh):

* HIV-1 infection documented by HIV ELISA and WB
* Age greater than or equal to 18 years old
* Hgb greater than or equal to 12 mg/dl
* CD4 greater than 200 cells/ micro liter and CD4% greater than 14% and not requiring prophylaxis for opportunistic infections
* Therapy with accepted HAART regimen for greater than or equal to 6 months.
* Viral load less than 50 copies RNA /ml plasma by RT-PCR for at least four months.
* Viral load greater than or equal to 0.38 copies RNA/ml plasma by SCA assay or positive in the adapted Amplicor assay
* Current HAART with DHHS-approved regimen NRTI+PI, NRTI alone, NRTI+NNRTI.
* Willingness to take an additional antiretroviral to current regimen for 30 days.
* For patients to start lopinavir/ritonavir, willingness to reduce the dose of sildenafil and other co-administered medicines that may be affected by the addition of lopinavir/ritonavir during the course of therapy with lopinavir/ritonavir
* For patients to start efavirenz arm, willingness to take efavirenz and adjust other medications or supplements as necessary, and to be aware that efavirenz is contraindicated in pregnancy and that may result in false positive urine tests for THC
* Patient must have primary care outside this protocol.
* Patients must practice accepted barrier methods to prevent pregnancy.

EXCLUSION CRITERIA:

* Requirement for cytotoxic agents including hydroxyurea or vaccinations during the study period
* Chronic corticosteroid therapy
* Concurrent therapy with investigational cytokines including IL-2 or IL-12 during the course of the study. Prior administration of cytokines is not an exclusion criteria; at least 4 months from most recent cycle of IL-2 or IL-12. GCSF and erythropoietin therapy will be permitted
* History of taking a salvage regimen; i.e., patient has had clinical resistance to antiretrovirals. Changing antiviral therapy because of adverse effects is permitted
* Prior PI therapy or NNRTI therapy is not permitted unless the previous PI-containing therapy was switched because of patient preference. If the patient has a documented history of lipid elevations (fasting triglycerides greater than 750 mg/dl), the patient will not be eligible for PI addition.
* Any febrile illness (T greater than 38.0 degrees C) in the 3 weeks prior to enrollment
* Any vaccination in the 6 weeks prior to enrollment
* Current pregnancy or lactation, history of pregnancy in the last 4 months
* Prior history of intolerance to the added antiretroviral
* For lopinavir/ritonavir addition, baseline elevated triglycerides greater than 400 mg/dl without lipid lowering agents
* Elevated baseline ALT liver function assays greater than 2 fold greater than upper limit of normal
* Known history of liver disease or Child-Pugh score greater than 5.
* History of pancreatitis requiring hospitalization
* Concomitant use with drugs that are highly dependent on cytochrome P450 for clearance, which, in the opinion of the investigators, may lead to the unexpected changes in their concentrations occurring after the addition of lopinavir/ritonavir or efavirenz. Examples include but are not limited to: wafarin-like anticoagulation , amiodarone, astemizole, cisapride, statin class of drugs, gemfibrozil, cyclosporine, ergonavine, ergotamine, methylergonavine, dihydroergotamine, dofetilide, flecanide, quinidine, fusidic acid, methadone, demerol, midazolam, triazolam, phenytoin, dilantin, pimozide, sirolimus, tacrolimus, propafenone, quinupristin, terfenadine, theophylline, rifampin, rifapentene, or rifabutin and illicit substances, including the recreational substance (ecstasy) methylenedioxymethamphetamine.
* History of chronic diarrhea or inflammatory bowel disease
* History of hemophilia
* Inability to comply with the protocol

For those starting efavirenz, significant depression, which, in the opinion of the investigators, would be significantly worsened by efavirenz.

INCLUSION CRITERIA - DRUG OVERLAP COHORT:

* HIV-1 infection documented by HIV ELISA and WB
* Age greater than or equal to18 years old
* Hgb greater than or equal to 12 mg/dl
* CD4 greater than 200 cells/ micro liter and CD4% greater than 14% and not requiring prophylaxis for opportunistic infections
* Therapy with accepted HAART regimen for greater than or equal to 6 months
* Viral load less than 50 copies RNA/ml plasma by RT-PCR for at least four months
* Viral load greater than 0.38 copies RNA/ml plasma by SCA assay or positive in the adapted Amplicor assay
* Current HAART with DHHS-approved regimen NRTI+PI, NRTI alone, NRTI+NNRTI
* Willingness to take an additional antiretroviral to current regimen for 30 days
* For patients planning to start lopinavir/ritonavir, or other ritonavir containing regimen willingness to reduce the dose of sildenafil and other co-administered medicines that may be affected by the addition of ritonavir during the course of therapy with lopinavir/ritonavir
* For patients to start efavirenz, willingness to take efavirenz and adjust other medications or supplements as necessary, and to be aware that efavirenz is contraindicated in pregnancy and that may result in false positive urine tests for THC
* Patient must have primary care outside this protocol
* Patients must practice accepted barrier methods to prevent pregnancy.

EXCLUSION CRITERIA:

* Requirement for cytotoxic agents including hydroxyurea or vaccinations during the study period
* Chronic corticosteroid therapy
* Concurrent therapy with investigational cytokines including IL-2 or IL-12 during the course of the study. Prior administration of cytokines is not an exclusion criteria; at least 4 months from most recent cycle of IL-2 or IL-12. GCSF and erythropoietin therapy will be permitted
* History of taking a salvage regimen; i.e., patient has had clinical resistance to antiretrovirals. Changing antiviral therapy because of adverse effects is permitted
* Prior PI therapy or NNRTI therapy is not permitted unless the previous PI-containing therapy was switched because of patient preference. If the patient has a documented history of lipid elevations (fasting triglycerides greater than 750 mg/dl) the patient will not be eligible for PI addition.
* Any febrile illness (T greater than 38 degrees C) in the 3 weeks prior to enrollment
* Any vaccination in the 6 weeks prior to enrollment
* Current Pregnancy or lactation, history of pregnancy in the last 4 months
* Prior history of intolerance to the added antiretroviral
* For protease addition, baseline elevated triglycerides greater than 400 mg/dl without lipid lowering agents
* Elevated baseline ALT liver function assays greater than 2 fold greater than upper limit of normal
* Known history of liver disease or Child-Pugh score greater than 5.
* History of pancreatitis requiring hospitalization
* For patients who are adding ritonavir or efavirenz, concomitant use with drugs that are highly dependent on cytochrome P 450 for clearance, which, in the opinion of the investigators, may lead to the unexpected changes in their concentrations occurring after the new drug is added. Examples include but are not limited to: wafarin-like anticoagulation , amiodarone, astemizole, cisapride, statin class of drugs, gemfibrozil, cyclosporine, ergonavine, ergotamine, methylergonavine, dihydroergotamine, dofetilide, flecanide, quinidine, fusidic acid, methadone, demerol, midazolam, triazolam, phenytoin, dilantin, pimozide, sirolimus, tacrolimus, propafenone, quinupristin, terfenadine, theophylline, rifampin, rifapentene, or rifabutin and illicit substances, including the recreational substance (ecstasy) methylenedioxymethamphetamine
* History of chronic diarrhea or inflammatory bowel disease
* History of hemophilia
* Inability to comply with the protocol
* For those starting efavirenz, significant depression, which, in the opinion of the investigators, would be significantly worsened by efavirenz

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2002-07-26; Study Completion 2013-02-07

CONTACTS AND LOCATIONS:
Overall Officials: Frank Maldarelli, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gallego O, Ruiz L, Vallejo A, Ferrer E, Rubio A, Clotet B, Leal M, Soriano V; ERASE-3 Group. Changes in the rate of genotypic resistance to antiretroviral drugs in Spain. AIDS. 2001 Sep 28;15(14):1894-6. doi: 10.1097/00002030-200109280-00025. PMID 11579258
- [Background] Lucas GM, Chaisson RE, Moore RD. Highly active antiretroviral therapy in a large urban clinic: risk factors for virologic failure and adverse drug reactions. Ann Intern Med. 1999 Jul 20;131(2):81-7. doi: 10.7326/0003-4819-131-2-199907200-00002. PMID 10419445
- [Background] Adje C, Cheingsong R, Roels TH, Maurice C, Djomand G, Verbiest W, Hertogs K, Larder B, Monga B, Peeters M, Eholie S, Bissagene E, Coulibaly M, Respess R, Wiktor SZ, Chorba T, Nkengasong JN; UNAIDS HIV Drug Access Initiative, Abidjan, Cote d'Ivoire. High prevalence of genotypic and phenotypic HIV-1 drug-resistant strains among patients receiving antiretroviral therapy in Abidjan, Cote d'Ivoire. J Acquir Immune Defic Syndr. 2001 Apr 15;26(5):501-6. doi: 10.1097/00126334-200104150-00018. PMID 11391173